CLINICAL TRIAL: NCT01821573
Title: Double Blind Randomized Controlled Study of the Effect of Botulinum Toxin Injection in Rectus Femoris and Triceps on the Length and the Strength of These Muscles During Locomotion in Chronic Hemiparetic Patients
Brief Title: Study of the Effect of Botulinum Toxin Injection in Rectus Femoris and Triceps on the Length and the Strength During Locomotion in Chronic Hemiparetic Patients
Acronym: FOLOTOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P110136 / AOM11223; 2012-001203-21 (EudraCT Number)
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-02

CONDITIONS: COMPARISON BETWEEN GROUP TREATED WITH BOTULINUM TOXIN AND PLACEBO
Keywords: botulinum toxin injection,3D motion analysis, muscular lengthening,muscle strength
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botox Injection (Experimental): Patients treated by botulinum toxin.
  Interventions: Drug: botulinum toxin type A
- Saline Solution (Placebo Comparator): Patients treated with saline solution.
  Interventions: Drug: injection of NaCl 0.9%

INTERVENTIONS:
Drug: botulinum toxin type A — Experimental arm group:
  * 150 Units in rectus femoris ( 3 ml and 3 points)
  * 70 units in medial gastrocnemius (1.4 ml and 1 point)
  * 70 units in lateral gastrocnemius ( 1.4 ml and 1 point)
  * 60 units in soleus ( 1.2 ml and 3 points)
  Other Names: Botox® allergan Inc
  Arms: Botox Injection
Drug: injection of NaCl 0.9% — Placebo comparator group: injection of NaCl 0.9%:
  * 3 ml of NaCl 0.9% in rectus femoris in 3 points
  * 1.4 ml of NaCl 0.9% in medial gastrocnemius in 1 point
  * 1.4 ml of Nacl 0.9% in lateral gastrocnemius in 1 point
  * 1.2 ml of NaCl 0.9% in soleus in 3 points
  Arms: Saline Solution

SUMMARY:
The aim of this randomized controlled study is to quantify the modification during locomotion of chronic hemiparetic patients of the strength and the length of Rectus Femoris and Triceps Surae induced by botulinum toxin injection type A.

The main hypotheses of this study based on previous studies are that botulinum toxin injection increases on one hand the length of the muscle injected during gait and on the other hand decreased the strength of the muscles injected.

The investigators also hypothesized that botulinum toxin injection improved the strength of the antagonist muscles and normalized the pattern of strength of the muscles injected during gait.

DETAILED DESCRIPTION:
The aim of this study is to compare versus placebo the effects of BTX-A injection on :

* the maximal length of the muscles injected during gait
* the maximal lengthening velocity of the muscles injected during gait
* the maximal strength of muscles injected during gait
* the inter-limb coordination assessed by continuous relative phase
* the kinematic parameters such as peak knee flexion during swing phase of the gait cycle and peak ankle dorsiflexion during stance phase.

To that end each patient included in the study will be assessed before injection, one month after the BTX-A injection and 3 months after BTX-A injections.

All patients will underwent a clinical examination, a 3D gait analysis and a isokinetic dynamometer analysis.

The comparison of the results in the group treated by BTX-A will permit to show that one month after BTX-A injection peak length during gait of muscles injected, maximal lengthening velocity peak knee flexion during swing phase and peak ankle dorsiflexion increase significantly.

It will also permit to show that the maximal strength of muscles injected decreases whereas the strength of antagonist increases It will also permit to demonstrate that multisite BTX-A injection improve coordination of paretic and non paretic lower limb the inter-group comparison will permit to demonstrate that these modification are mainly due to multisite BTX-A injections.

ELIGIBILITY:
Inclusion Criteria:

* men or women aged > 18 ans
* unilateral stroke more than 6 months
* ability to walk 10 meters without assistive device
* decrease of peak knee flexion in swing phase of the gait cycle due to a spasticity of Rectus femoris muscle
* plantarflexion in swing phase of the gait cycle due to a spasticity of the triceps surae
* informed consent approved
* oral contraception

Exclusion Criteria:

* Aphasia
* anteriority of lower limb surgery less than 6 months
* underlying disease
* pre-existing neuro-muscular disorders
* pregnancy
* absence of oral contraception
* last botulinum toxin injection < 3months
* hypersensitivity reactions
* co-administration of aminoglycosides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Measure of the maximal length of the muscles treated by Botulinum | 1.5 hours
  The maximal length of the muscles treated by Botulinum Toxin during locomotion quantified using 3D motion analysis and musculo-skeletal model.
  This measure will be performed one month after Botulinum toxin injection.

SECONDARY OUTCOMES:
The maximal strength measure | 1.5 hours
  The maximal strength developed by injected muscles during gait.
Inter-segmental coordination measure | 1.5 hours
  The modification of inter-segmental coordination during locomotion induced by botulinum toxin and quantified by continuous relative phase injection
Measure of joint torque at knee and ankle level. | 1.5 hours
  The modification of joint torque at knee and ankle level induced by botulinum toxin injection.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Roche, MD, Principal Investigator — Physical medicine and rehabilation Department, Hôpital RAYMOND POINCARE, 92380 Garches, France
Locations (3):
- France (3):
  - Service de médecine physique et réadaptation CHU de Brest, Brest, Brittany Region
  - Nicolas Roche, Garches, Hauts-de-Seine
  - Centre de rééducation de l'ADAPT Montargis, Amilly, Loiret

REFERENCES:
- [Derived] Supiot A, Geiger M, Bensmail D, Aegerter P, Pradon D, Roche N. Effect of botulinum toxin injection on length and force of the rectus femoris and triceps surae muscles during locomotion in patients with chronic hemiparesis (FOLOTOX). BMC Neurol. 2018 Aug 2;18(1):104. doi: 10.1186/s12883-018-1110-8. PMID 30068305